CLINICAL TRIAL: NCT03670862
Title: Prediction Model for the Recanalization Outcome Evaluation of Ischemic Stroke Using Multimodal CT
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: PROTECT-ChinaPLAGH
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Stroke, Acute
Keywords: Ischemic stroke; CTP; CTA
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke: Ischemic stroke patients with sympton onset in 24 hours
  Interventions: Other: CT

INTERVENTIONS:
Other: CT — Non-contrast computed tomography , computed tomography angiography, computed tomography perfusion imaging

SUMMARY:
Prediction model for the Recanalization OuTcome Evaluation of ischemic stroke using multimodal CT (PROTECT) study was a multicenter prospective observational study that recruited patients from 13 centers located in 10 provinces across China. The study was to assess the effects of novel imaging biomarkers/ imaging patterns based on multimodel CT for patients selection and outcome prediction in acute ischemic stroke.

DETAILED DESCRIPTION:
Patients Patients with cerebral ischemia symptoms of anterior circulation or posterior circulation onset in 24 hours were included. A neurological evaluation (Modified Rankin Scale and NIHSS); physical examination, including measurement of weight (kg) and vital signs (supine systolic and diastolic blood pressure); time from symptom onset to enrollment were recorded.

Imaging protocols:

CT scan protocols: Non-contrast computed tomography(NCCT) , computed tomography angiography(CTA), computed tomography perfusion(CTP)

Contrast agent:

CTA: Omniscan 40-50ml, 5ml/s; saline solution 50ml, 5ml/s

CTP: Omniscan 50ml, 5ml/s; saline solution 50ml, 5ml/s

Imaging evaluation:

CTA was reviewed and stenosis or occlusive lesions were identified. Parameter maps including cerebral blood flow, cerebral blood volume, mean transit time, the time to the maximum of the residue function derived from CTP were processed by the software Rapid to quantitatively assess infarct core volume and mismatch.

Multiphase CTA was extracted from CTP to evaluate the collateral circulation.

Treatment:

Intravenous recombinant tissue plasminogen activator(rtPA), endovascular therapy, and conventional treatment including neuroprotection, anti-platelet, and statin according to the guideline.

Follow up:

Modified Rankin Scale(mRS) was obtained at 90 days after symptom onset. An imaging follow-up was also recommended within 30 days after symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral ischemic sympton with onset in 24 hours
* All CT examination performed according to study protocol
* Signed informed consent obtained from the patient or patient's legally authorized representative

Exclusion Criteria:

* Acute intracranial hemorrhage
* Pre-existing medical, the neurological, or psychiatric disease that would confound the neurological, functional, or imaging evaluations
* Pregnancy
* Known allergy to iodine previously refractory to pretreatment medications
* Renal Failure (serum creatinine > 2.0 or Glomerular Filtration Rate < 30)
* History of severe kidney disease as an adult, including tumor or transplant surgery, or family history of kidney failure
* Severe cardiac insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients with sympton onset in 24 hours
Sampling Method: Probability Sample
Enrollment: 862 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
90-day functional outcome | 90 days after symptom onset
  Assessed by modified Rankin Scale with scores ranging from 0 (no symptoms) to 6 (death)

SECONDARY OUTCOMES:
Final infarction volume | within 30 days after symptom onset
  Finding the predictive value of novel imaging biomarkers/ imaging patterns on final infarction volume
Percentage of Hemorrhagic Transformation | within 7 days after symptom onset
  Symptomatic hemorrhagic transformation after acute ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, M.D.,Ph.D., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China